CLINICAL TRIAL: NCT06267001
Title: A Phase III, Randomized, Double-blind Study of Tiragolumab Plus Atezolizumab Compared With Placebo Plus Atezolizumab in Participants With Completely Resected Stage IIB, IIIA, or Select IIIB, PD-L1 Positive, Non-small Cell Lung Cancer Who Have Received Adjuvant Platinum-based Chemotherapy
Brief Title: A Study of Tiragolumab Plus Atezolizumab Compared With Placebo Plus Atezolizumab in Participants With Completely Resected Non-small Cell Lung Cancer Who Have Received Adjuvant Platinum-based Chemotherapy
Acronym: SKYSCRAPER-15
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO45006; 2023-506696-10-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Tiragolumab (Experimental): Participants will receive atezolizumab and tiragolumab intravenously (IV).
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Atezolizumab + Placebo (Placebo Comparator): Participants will receive atezolizumab and placebo IV.
  Interventions: Drug: Atezolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered IV.
  Other Names: Tecentriq; RO5541267
Drug: Tiragolumab — Tiragolumab will be administered IV.
  Other Names: MTIG7192A; RO7092284
  Arms: Atezolizumab + Tiragolumab
Drug: Placebo — Placebo will be administered IV.
  Arms: Atezolizumab + Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of tiragolumab plus atezolizumab compared with placebo plus atezolizumab administered to participants with non-small cell lung cancer (NSCLC) following resection and adjuvant chemotherapy.

DETAILED DESCRIPTION:
With Protocol Amendment 2, enrollment will be stopped. The primary objective of the study has been changed to a safety objective and no other analysis will be conducted

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histological or cytological diagnosis of Stage IIB, IIIA, and select IIIB NSCLC of either non-squamous or squamous histology
* Participants must have had complete resection of NSCLC
* Participants must have received between one to four cycles of adjuvant histology-based platinum doublet chemotherapy
* Participants must have recovered adequately from surgery and from adjuvant chemotherapy
* Tumor cell PD-L1 expression at >/= 1%
* Adequate hematologic and end-organ function.

Exclusion Criteria:

* Any history of prior NSCLC within the last 5 years
* Any evidence of residual disease or disease recurrence following surgical resection of NSCLC, or during or following adjuvant chemotherapy
* NSCLC known to have mutation in the epidermal growth factor receptor (EGFR) gene or an anaplastic lymphoma kinase (ALK) fusion oncogene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- Centro Oncologico Korben, Ciudad Autonoma Buenos Aires, Argentina
- Australia (2):
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Monash Health, Clayton, Victoria
- Brazil (6):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Nucleo de Oncologia da Bahia - NOB, Salvador, Bahia, Estado de Bahia
  - Hospital de Clínicas de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital A. C. Camargo, São Paulo, São Paulo
- China (11):
  - Changzhou First People's Hospital, Changzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Shandong Cancer Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Ningbo No.2 Hospital, Ningbo
  - Liaoning Provincial Cancer Hospital, Shengyang
  - Tianjin Cancer Hospital, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Zhejiang Cancer Hospital, Zhejiang
- Ospedale P. Pederzoli Casa di cura Privata, Peschiera Del Garda (VR), Veneto, Italy
- Japan (2):
  - Hiroshima University Hospital, Hiroshima
  - Kindai University Hospital, Osaka
- Instytut Gruzlicy I Chorob Pluc, Warsaw, Poland
- South Korea (10):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - St. Vincent's Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Taiwan (3):
  - E-DA Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Cancer Center, Zhongzheng Dist.
- Vajira Hospital, Bangkok, Thailand
- Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Tibbi Onkoloji, Bakirkoy / Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing
Access Criteria: Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).